CLINICAL TRIAL: NCT03651700
Title: A Phase II, Randomized Blinded Study of the Effects of Transcranial Magnetic Stimulation and Constraint Induced Language Therapy for the Treatment of Chronic Aphasia
Brief Title: Transcranial Magnetic Stimulation and Constraint Induced Language Therapy for Chronic Aphasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Branch Coslett (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, H. Branch Coslett, Professor, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 831532-chbdfejh; R01DC016800 (NIH)
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either TMS or sham TMS in a 2:1 allocation ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The individual administering TMS will keep the master file of subject assignments, but all other individuals in contact with the subject or their data will be unaware of group assignment. Participants will not be informed of their assignment to active or sham status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TMS (Active Comparator): There will be 10 TMS sessions over 2 consecutive weeks in which 20 minutes (1200 pulses) of 1 Hz active TMS will be delivered to the inferior pars triangular. Each TMS treatment session will be immediately followed by a 60-90 minute session of Constrained Induced Language Therapy (CILT).
  Interventions: Device: Active TMS; Behavioral: CILT
- Sham TMS (Sham Comparator): There will be 10 TMS sessions over 2 consecutive weeks in which 20 minutes (1200 pulses) of 1 Hz sham TMS will be delivered to the inferior pars triangular. Sham TMS will be administered with a sham TMS coil that looks and sounds like the active coil but does not generate a magnetic field. Each TMS treatment session will be immediately followed by a 60-90 minute session of Constrained Induced Language Therapy (CILT).
  Interventions: Device: Sham TMS; Behavioral: CILT

INTERVENTIONS:
Device: Active TMS — Active TMS will be at 90% motor threshold
  Arms: Active TMS
Device: Sham TMS — Sham TMS will be administered
  Arms: Sham TMS
Behavioral: CILT — 60-90 minutes of CILT will be administered during each treatment session
  Other Names: Constraint Induced Language Therapy

SUMMARY:
Transcranial Magnetic Stimulation (TMS) has been demonstrated to improve language function in subjects with chronic aphasia in a number of small studies, many of which did not include a control group. Although the treatment appears promising, data to date do not permit an adequate assessment of the utility of the technique. The investigators propose to study the effects of TMS combined with Constraint Induced Language Therapy (CILT) in 75 subjects with chronic aphasia. Subjects will be randomized in a 2:1 ratio to TMS with CILT or sham TMS with CILT. One Hz TMS at 90% motor threshold will be delivered to the right inferior frontal gyrus for 20 minutes in 10 sessions over 2 weeks; language therapy will be provided for one hour immediately after the conclusion of each session of TMS. Change from baseline in the Western Aphasia Battery Aphasia Quotient at 6 months after the end of TMS treatment will serve as the primary outcome measure.

DETAILED DESCRIPTION:
TMS is a technique by which a brief electrical current is induced in brain tissue causing a brief suppression of the excitability of the underlying tissue; the technique, which was introduced in the 1980s and has been extensively used around the world, has been shown to transiently improve or disrupt specific cognitive operations. To achieve this end, a coil is positioned against the subject's head. The delivery of a single pulse begins with the discharge of current from a capacitor into a circular or figure-of-eight coil; this electrical current generates a brief magnetic field of up to 2.2 Tesla. As the pulse of electricity has a rise time of 0.2 ms. and a duration of 1 ms., the magnetic field changes in intensity quite rapidly. Because the magnetic field passes freely through the scalp, skull, and meninges, the flux in the magnetic field induces a small electric field in the brain that transiently alters neural activity.

TMS may be delivered in a variety of ways. The investigators propose to use 1 Hz TMS; that is, TMS pulses will be delivered at a frequency of 1/second. This style of TMS is assumed to be inhibitory in that it transiently suppresses the function of the cortex under the coil. Using the figure-of-eight coil to be employed here, TMS is thought to reduce activity in approximately 1 cubic cm. of cortex. Many investigators have employed TMS with a frequency of 1 Hz for periods of 20 minutes and longer; mild behavioral deficits are often present for several minutes in these studies.

The baseline phase will consist of 3 sessions, each lasting 1-2 hours depending on the stamina of the subject. The point of the baseline testing is to characterize the subject's language function. To that end, a number of standard language and neuropsychological tasks will be administered. These include the Western Aphasia Battery, Pyramids and Palm Trees test, Figural Fluency Test, word and non-word repetition tasks, the Nicholas and Brookshire Narratives, CILT stimulus naming, and Northwestern Assessment of Verbs and Sentences. Additionally, during the baseline, subjects will undergo MRI of the brain or, if they have a contraindication to MRI, a CAT scan of the head. No contrast will be used.

In the treatment phase, there will be 10 TMS sessions over 2 consecutive weeks in which 20 minutes (1200 pulses) of 1 Hz TMS at 90% motor threshold will be delivered to the inferior pars triangularis. Each TMS treatment session will be immediately followed by a 60-90 minute session of CILT

There will be two 3-month post-treatment visits and two 6-month post-treatment visits in which the full battery of language and cognitive assessments will be repeated. Subjects who are able to undergo MRI scanning will have anatomic and fMRI scans at the first 6-month post-treatment visit.

The investigators will pair TMS with CILT which has been shown to have positive outcomes in post-stroke aphasia. CILT invokes use-dependent learning in communicative interactions by requiring spoken output and restricting use of alternative forms of communication, such as gestures. The investigators will use a dual card-matching task modeled after Maher et al. As in the original CILT design, the participant interacts verbally with a conversational partner (here, the speech language pathologist), in turn requesting a card of given description and complying with the partner's request. In this way, the treatment targets both production and comprehension. Moreover, as verbal targets increase in linguistic complexity across the protocol ("a ball", "throw a ball"; "Do you have a ball"?), a variety of lexical and phrasal structures are targeted. Studies of CILT have reported gains on multiple language behaviors, supporting its broad engagement of the language network.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence and MRI or CT verification of a single left hemisphere stroke with moderate to severe aphasia.
* Suffered their stroke at least 6 months prior to their testing
* Must be able to understand the nature of the study, and give informed consent

Exclusion Criteria:

* Multiple strokes (excluding small lacunar strokes) as defined by brain imaging
* History of substance abuse
* Previous head trauma with loss of consciousness for more than 5 minutes
* Psychiatric illness (We note that subjects will be assessed with the 15-item Geriatric Depression scale. Because depression is very difficult to evaluate in aphasic subjects, potential subjects will not be excluded on the basis of the depression score)
* Chronic exposure to medications that might be expected to have lasting consequences for the central nervous system (e.g. haloperidol, dopaminergics)
* History of or neuropsychological findings suggestive of dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Branch Coslett, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shewan CM, Kertesz A. Reliability and validity characteristics of the Western Aphasia Battery (WAB). J Speech Hear Disord. 1980 Aug;45(3):308-24. doi: 10.1044/jshd.4503.308. PMID 7412225
- [Background] Howard, D., & Patterson, K. E. (1992). The Pyramids and Palm Trees Test: A Test of Semantic Access from Words and Pictures. Thames Valley Test Company. Retrieved from books.google.com/books?id=dykONQAACAAJ
- [Background] Ruff, R. M. (1996). Ruff figural fluency test: professional manual. Psychological Assessment Resources.
- [Background] Nicholas LE, Brookshire RH. A system for quantifying the informativeness and efficiency of the connected speech of adults with aphasia. J Speech Hear Res. 1993 Apr;36(2):338-50. doi: 10.1044/jshr.3602.338. PMID 8487525
- [Background] Pulvermuller F, Neininger B, Elbert T, Mohr B, Rockstroh B, Koebbel P, Taub E. Constraint-induced therapy of chronic aphasia after stroke. Stroke. 2001 Jul;32(7):1621-6. doi: 10.1161/01.str.32.7.1621. PMID 11441210
- [Background] Maher LM, Kendall D, Swearengin JA, Rodriguez A, Leon SA, Pingel K, Holland A, Rothi LJ. A pilot study of use-dependent learning in the context of Constraint Induced Language Therapy. J Int Neuropsychol Soc. 2006 Nov;12(6):843-52. doi: 10.1017/S1355617706061029. PMID 17064447
- [Background] Barthel, G., Meinzer, M., Djundja, D., & Rockstroh, B. (2008). Intensive language therapy in chronic aphasia: Which aspects contribute most? Aphasiology, 22(4), 408-421.
- [Background] Goral M, Kempler D. TRAINING VERB PRODUCTION IN COMMUNICATIVE CONTEXT: EVIDENCE FROM A PERSON WITH CHRONIC NON-FLUENT APHASIA. Aphasiology. 2009 Dec 12;23(12):1383-1397. doi: 10.1080/02687030802235203. PMID 19911035
- [Background] Meinzer M, Rodriguez AD, Gonzalez Rothi LJ. First decade of research on constrained-induced treatment approaches for aphasia rehabilitation. Arch Phys Med Rehabil. 2012 Jan;93(1 Suppl):S35-45. doi: 10.1016/j.apmr.2011.06.040. PMID 22202189
- [Background] Abo M, Kakuda W, Watanabe M, Morooka A, Kawakami K, Senoo A. Effectiveness of low-frequency rTMS and intensive speech therapy in poststroke patients with aphasia: a pilot study based on evaluation by fMRI in relation to type of aphasia. Eur Neurol. 2012;68(4):199-208. doi: 10.1159/000338773. Epub 2012 Aug 29. PMID 22948550
- [Background] Avenanti A, Coccia M, Ladavas E, Provinciali L, Ceravolo MG. Low-frequency rTMS promotes use-dependent motor plasticity in chronic stroke: a randomized trial. Neurology. 2012 Jan 24;78(4):256-64. doi: 10.1212/WNL.0b013e3182436558. Epub 2012 Jan 11. PMID 22238412
- [Background] Barwood CH, Murdoch BE, Riek S, O'Sullivan JD, Wong A, Lloyd D, Coulthard A. Long term language recovery subsequent to low frequency rTMS in chronic non-fluent aphasia. NeuroRehabilitation. 2013;32(4):915-28. doi: 10.3233/NRE-130915. PMID 23867417
- [Background] Barwood CHS, Murdoch BE, Whelan BM, Lloyd D, Riek S, O'Sullivan JD, Coulthard A, Wong A. Improved receptive and expressive language abilities in nonfluent aphasic stroke patients after application of rTMS: an open protocol case series. Brain Stimul. 2012 Jul;5(3):274-286. doi: 10.1016/j.brs.2011.03.005. Epub 2011 Apr 13. PMID 22037124
- [Background] Hamilton RH, Sanders L, Benson J, Faseyitan O, Norise C, Naeser M, Martin P, Coslett HB. Stimulating conversation: enhancement of elicited propositional speech in a patient with chronic non-fluent aphasia following transcranial magnetic stimulation. Brain Lang. 2010 Apr;113(1):45-50. doi: 10.1016/j.bandl.2010.01.001. Epub 2010 Feb 16. PMID 20159655
- [Background] Hara T, Abo M, Kobayashi K, Watanabe M, Kakuda W, Senoo A. Effects of low-frequency repetitive transcranial magnetic stimulation combined with intensive speech therapy on cerebral blood flow in post-stroke aphasia. Transl Stroke Res. 2015 Oct;6(5):365-74. doi: 10.1007/s12975-015-0417-7. Epub 2015 Aug 7. PMID 26245774
- [Background] Kakuda W, Abo M, Momosaki R, Morooka A. Therapeutic application of 6-Hz-primed low-frequency rTMS combined with intensive speech therapy for post-stroke aphasia. Brain Inj. 2011;25(12):1242-8. doi: 10.3109/02699052.2011.608212. Epub 2011 Sep 8. PMID 21902549
- [Background] Kakuda W, Abo M, Shimizu M, Sasanuma J, Okamoto T, Yokoi A, Taguchi K, Mitani S, Harashima H, Urushidani N, Urashima M; NEURO Investigators. A multi-center study on low-frequency rTMS combined with intensive occupational therapy for upper limb hemiparesis in post-stroke patients. J Neuroeng Rehabil. 2012 Jan 20;9(1):4. doi: 10.1186/1743-0003-9-4. PMID 22264239
- [Background] Kakuda W, Abo M, Uruma G, Kaito N, Watanabe M. Low-frequency rTMS with language therapy over a 3-month period for sensory-dominant aphasia: case series of two post-stroke Japanese patients. Brain Inj. 2010;24(9):1113-7. doi: 10.3109/02699052.2010.494587. PMID 20569046
- [Background] Khedr EM, Abo El-Fetoh N, Ali AM, El-Hammady DH, Khalifa H, Atta H, Karim AA. Dual-hemisphere repetitive transcranial magnetic stimulation for rehabilitation of poststroke aphasia: a randomized, double-blind clinical trial. Neurorehabil Neural Repair. 2014 Oct;28(8):740-50. doi: 10.1177/1545968314521009. Epub 2014 Feb 6. PMID 24503205
- [Background] Kindler J, Schumacher R, Cazzoli D, Gutbrod K, Koenig M, Nyffeler T, Dierks T, Muri RM. Theta burst stimulation over the right Broca's homologue induces improvement of naming in aphasic patients. Stroke. 2012 Aug;43(8):2175-9. doi: 10.1161/STROKEAHA.111.647503. Epub 2012 May 10. PMID 22581821
- [Background] Martin PI, Naeser MA, Ho M, Treglia E, Kaplan E, Baker EH, Pascual-Leone A. Research with transcranial magnetic stimulation in the treatment of aphasia. Curr Neurol Neurosci Rep. 2009 Nov;9(6):451-8. doi: 10.1007/s11910-009-0067-9. PMID 19818232
- [Background] Martin PI, Naeser MA, Theoret H, Tormos JM, Nicholas M, Kurland J, Fregni F, Seekins H, Doron K, Pascual-Leone A. Transcranial magnetic stimulation as a complementary treatment for aphasia. Semin Speech Lang. 2004 May;25(2):181-91. doi: 10.1055/s-2004-825654. PMID 15118944
- [Background] Martin PI, Treglia E, Naeser MA, Ho MD, Baker EH, Martin EG, Bashir S, Pascual-Leone A. Language improvements after TMS plus modified CILT: Pilot, open-protocol study with two, chronic nonfluent aphasia cases. Restor Neurol Neurosci. 2014;32(4):483-505. doi: 10.3233/RNN-130365. PMID 25015701
- [Background] Medina J, Norise C, Faseyitan O, Coslett HB, Turkeltaub PE, Hamilton RH. Finding the Right Words: Transcranial Magnetic Stimulation Improves Discourse Productivity in Non-fluent Aphasia After Stroke. Aphasiology. 2012 Sep 1;26(9):1153-1168. doi: 10.1080/02687038.2012.710316. Epub 2012 Aug 29. PMID 23280015
- [Background] Naeser MA, Martin PI, Lundgren K, Klein R, Kaplan J, Treglia E, Ho M, Nicholas M, Alonso M, Pascual-Leone A. Improved language in a chronic nonfluent aphasia patient after treatment with CPAP and TMS. Cogn Behav Neurol. 2010 Mar;23(1):29-38. doi: 10.1097/WNN.0b013e3181bf2d20. PMID 20299861
- [Background] Naeser MA, Martin PI, Nicholas M, Baker EH, Seekins H, Helm-Estabrooks N, Cayer-Meade C, Kobayashi M, Theoret H, Fregni F, Tormos JM, Kurland J, Doron KW, Pascual-Leone A. Improved naming after TMS treatments in a chronic, global aphasia patient--case report. Neurocase. 2005 Jun;11(3):182-93. doi: 10.1080/13554790590944663. PMID 16006338
- [Background] Naeser MA, Martin PI, Nicholas M, Baker EH, Seekins H, Kobayashi M, Theoret H, Fregni F, Maria-Tormos J, Kurland J, Doron KW, Pascual-Leone A. Improved picture naming in chronic aphasia after TMS to part of right Broca's area: an open-protocol study. Brain Lang. 2005 Apr;93(1):95-105. doi: 10.1016/j.bandl.2004.08.004. PMID 15766771
- [Background] Naeser MA, Martin PI, Theoret H, Kobayashi M, Fregni F, Nicholas M, Tormos JM, Steven MS, Baker EH, Pascual-Leone A. TMS suppression of right pars triangularis, but not pars opercularis, improves naming in aphasia. Brain Lang. 2011 Dec;119(3):206-13. doi: 10.1016/j.bandl.2011.07.005. Epub 2011 Aug 23. PMID 21864891
- [Background] Seniow J, Waldowski K, Lesniak M, Iwanski S, Czepiel W, Czlonkowska A. Transcranial magnetic stimulation combined with speech and language training in early aphasia rehabilitation: a randomized double-blind controlled pilot study. Top Stroke Rehabil. 2013 May-Jun;20(3):250-61. doi: 10.1310/tsr2003-250. PMID 23841973
- [Background] Szaflarski JP, Vannest J, Wu SW, DiFrancesco MW, Banks C, Gilbert DL. Excitatory repetitive transcranial magnetic stimulation induces improvements in chronic post-stroke aphasia. Med Sci Monit. 2011 Feb 25;17(3):CR132-9. doi: 10.12659/msm.881446. PMID 21358599
- [Background] Thiel A, Hartmann A, Rubi-Fessen I, Anglade C, Kracht L, Weiduschat N, Kessler J, Rommel T, Heiss WD. Effects of noninvasive brain stimulation on language networks and recovery in early poststroke aphasia. Stroke. 2013 Aug;44(8):2240-6. doi: 10.1161/STROKEAHA.111.000574. Epub 2013 Jun 27. PMID 23813984
- [Background] Waldowski K, Seniow J, Lesniak M, Iwanski S, Czlonkowska A. Effect of low-frequency repetitive transcranial magnetic stimulation on naming abilities in early-stroke aphasic patients: a prospective, randomized, double-blind sham-controlled study. ScientificWorldJournal. 2012;2012:518568. doi: 10.1100/2012/518568. Epub 2012 Nov 20. PMID 23213288
- [Background] Weiduschat N, Thiel A, Rubi-Fessen I, Hartmann A, Kessler J, Merl P, Kracht L, Rommel T, Heiss WD. Effects of repetitive transcranial magnetic stimulation in aphasic stroke: a randomized controlled pilot study. Stroke. 2011 Feb;42(2):409-15. doi: 10.1161/STROKEAHA.110.597864. Epub 2010 Dec 16. PMID 21164121

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2019-2024 from the Hospital of the University of Pennsylvania, surrounding Philadelphia area medical centers and aphasia support groups.
Pre-assignment Details: A total of 36 participants did not qualify due to medical contraindications (14) or aphasia severity (22).
  Nine participants dropped out of the study prior to randomization due to safety concerns (1), inability to complete MRI scan (3), lost to follow-up (2), travel concerns (1), no longer interested in participating (2).
Groups:
- Active TMS: Participants will receive 10 TMS sessions over 2 consecutive weeks in which 20 minutes (1200 pulses) of 1 Hz active TMS will be delivered to the inferior pars triangular.
  Each TMS treatment session will be immediately followed by a 60-90 minute session of Constrained Induced Language Therapy (CILT).
  Active TMS: Active TMS will be at 90% motor threshold
  CILT: 60-90 minutes of CILT will be administered during each treatment session
- Sham TMS: Participants will take part in 10 Sham TMS sessions over 2 consecutive weeks for 20 minutes each day. Sham TMS mimics the sensory experience (look, sound and feel) of active TMS but does not stimulate the brain. Sham TMS will be administered with a sham TMS coil that looks and sounds like the active coil but does not generate a magnetic field. The sham TMS will target the same brain location - left inferior pars triangularis.
  Each sham TMS treatment session will be immediately followed by a 60-90 minute session of Constrained Induced Language Therapy (CILT).
Period: Overall Study
Arm/Group | Active TMS | Sham TMS
Started | 26 | 15
Completed | 25 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS | Sham TMS | Total
Number analyzed (Participants) | 26 | 15 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.73 (10.62) | 61.67 (10.87) | 59.17 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 4 | 17
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 0 | 22
  Not Hispanic or Latino | 3 | 13 | 16
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 18 | 9 | 27
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Western Aphasia Battery (WAB-AQ) Score [Mean (Standard Deviation); unit: score on a scale] | 66.6 (19.9) | 68.8 (18.5) | 67.4 (18.7)
Philadelphia Naming Test, Items Correct [Mean (Standard Deviation); unit: number of items correct] | 110.4 (57.0) | 114.0 (42.6) | 111.7 (51.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in WAB-AQ
Description: The primary outcome measure will be the change in score on the Western Aphasia Battery Aphasia Quotient (WAB-AQ), a score assessing overall aphasia recovery. Scores can range from 0-100, with higher scores representing better outcomes. 0-25 is very severe, 26-50 is severe, 51-75 is moderate, and 76-above is mild. A score of 93 or higher is considered recovered.
Time Frame: 6-months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 25 | 15
score on a scale | 3.0 (3.8) | 2.8 (5.9)
Statistical Analysis 1: Comparison: Active TMS vs Sham TMS; Test type: Superiority; p < .05, t-test, 2 sided

2. Secondary Outcome: Change in Percentage of Items Correct on the PNT
Description: The secondary outcome measure will be change in naming accuracy on the Philadelphia Naming Test (PNT). PNT naming accuracy is measured as a percentage from 0% to 100% with higher percentages meaning better naming ability. The task involves naming 175 pictures of common objects.
Time Frame: 6-months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 25 | 15
score on a scale | 3.4 (8.9) | 3.4 (9.1)
Statistical Analysis 1: Comparison: Active TMS vs Sham TMS; Test type: Superiority; p < .05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From baseline, adverse event data were collected over a period of time consisting of 6 months.
Description: Adverse event (AEs) information was collected daily during treatment sessions, as well as each follow-up visit.
Arm/Group | Active TMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/15
Other Adverse Events (participants affected / at risk) | 13/26 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS (N=26) | Sham TMS (N=15)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — Generalized seizure occurred approximately 5 weeks after completion of treatment. Our DSMB agreed that this SAE was unrelated to the study.
Cancer Diagnosis (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS (N=26) | Sham TMS (N=15)
Cut/Wound Care (Infections and infestations) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 6 (6) | 1 (3)
Bladder Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Stiff Neck (General disorders) | 1 (1) | 1 (2)
Anxiety Attach (Psychiatric disorders) | 1 (1) | 0 (0)
Jaw Pain (General disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (2)
Atrial Fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0)
Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 1 (1) | 1 (1)
Facial Tingling (Nervous system disorders) | 1 (1) | 0 (0)
Broken Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1)
Nosebleed (General disorders) | 0 (0) | 1 (1)
Macular Edema (Eye disorders) | 0 (0) | 1 (1)
Vagus Nerve Stimulator (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT03651700/Prot_SAP_000.pdf